CLINICAL TRIAL: NCT05156385
Title: Sexual Dysfunction in Hypertensive Women According to Drug Adherence: Multicenter Cross-sectional Study
Brief Title: Sexual Dysfunction in Hypertensive Women
Acronym: DYSFHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/19/0553
Record Dates: First submitted 2021-10-15; First posted 2021-12-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
Keywords: high blood pressure; antihypertensive drugs; sexual dysfunction
MeSH Terms: conditions — Hypertension; Sexual Dysfunction, Physiological | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertensive women (Experimental)
  Interventions: Biological: Blood sample for the determination of antihypertensives or their metabolites.; Behavioral: Questionnaire on sexual activity; Behavioral: Scale on hospital anxiety and depression; Behavioral: Morisky Questionaire

INTERVENTIONS:
Biological: Blood sample for the determination of antihypertensives or their metabolites. — 15 ml of Blood sample for the determination of antihypertensives or their metabolites
Behavioral: Questionnaire on sexual activity — Questionnaire on sexual activity in women
Behavioral: Scale on hospital anxiety and depression — Scale on hospital anxiety and depression to detect anxious and depressive symptoms (14 questions)
Behavioral: Morisky Questionaire — anti-hypertensive medication compliance questionnaire

SUMMARY:
Several studies describe the existence of an association between sexual dysfunction and high blood pressure (hypertension), most often characterized by a decrease in the number of orgasms and the existence of dyspareunia.

Hypertension is a contributing factor, and nonadherence to medication could amplify it.

There are several ways to assess adherence to treatment: the use of declarative questionnaires, a method not without criticism because it is subject to the subjectivity of the declaration by the patient; and drug dosages, a standard technique, although insufficiently disseminated due to the high cost and greater weight of the survey protocols. Drug non-compliance is multifactorial. In addition, it has been shown that having undesirable drug effects and / or being afraid of developing them is one of the major causes of non-compliance with antihypertensive treatments.

The investigators hypothesize that DS is significantly more common among hypertensive women treated with non-observers compared to hypertensive women treated with observers.

The main objective is to compare the prevalence of sexual dysfunction between a group of hypertensive women treated as observers and a group of hypertensive women treated as non-observers.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18,
* Hospitalized or received in consultation for the management of hypertension treated in one of the hypertension and therapeutic, nephrology or cardiology departments participating in the study, with confirmed hypertension, treated with the following dosable antihypertensive agent(s): diltiazem, verapamil, acebutolol, atenolol, nébivolol, bisoprolol, metoprolol, propranolol, amiloride, furosemide, hydrochlorothiazide, indapamide, spironolactone, spironolactone, Lorsartan, Irbesartan, Ramipril, Perindopril, Amlodipine,
* Having signed the informed consent form.
* Beneficiary or affiliated to a French Social insurance

Exclusion Criteria:

* Patients with bariatric surgery,
* Patients under guardianship/trusteeship/protection of justice,
* Patients with diagnosed and treated psychosis or depression, - Pregnant or nursing women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Analyse of sexual dysfunction | 25 months
  Prevalence of sexual dysfunction defined by a score less than 26 on the Female Sexual Function Index scale : score less than 26 mean a sexual dysfunction

SECONDARY OUTCOMES:
Percentage of patients with a good medication compliance by drug dosages and the Morisky questionnaire | 25 months
  Compare two methods of assessing drug compliance: drug dosages in the blood and the Morisky questionnaire; The score is rated on 8 points. A score of 8 is considered "good observant", a score between 6 and 7 "moderately observant patient" and a score strictly lower than 6 "poor observant".
Number of cases with sexual dysfunction in hypertensive women according to the antihypertensive pharmacological classes used | 25 months
  Estimate the prevalence of sexual dysfunction according to the antihypertensive pharmacological classes used (in the biologicale analysis)
Number of cases with sexual dysfunction in hypertensive women according to the number of antihypertensive treatments; | 25 months
  Estimate the prevalence of sexual dysfunction according to the number of antihypertensive treatments;

CONTACTS AND LOCATIONS:
Overall Officials: Delphine LAZARO-VERGE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- LAZARO Delphine, Toulouse, CHU de Toulouse, France

IPD SHARING:
Plan to Share IPD: No